CLINICAL TRIAL: NCT01596153
Title: Randomized Double-blind, Placebo-Controlled Trial Comparing the the Effect of Enhance Probiotic (EP, Go Live Rx,) Versus Placebo (Pl) on the Incidence of Clostridium Difficile Associated Diarrhea (CDAD) or Antibiotic-Associated Diarrhea (AAD)in Hospitalized Patients Initiated on Antibiotics
Brief Title: Probiotics in Hospitalized Patients Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was not initiated
Sponsor: South Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: SSH 10-006
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-11

CONDITIONS: Antibiotic Associated Diarrhea; Clostridium Difficile Associated Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): BID
  Interventions: Dietary Supplement: Go Live
- Go Live Rx Probiotic (Active Comparator): BID
  Interventions: Dietary Supplement: Go Live

INTERVENTIONS:
Dietary Supplement: Go Live — Enhanced Probiotic, one packet bid until 7 days after discontinuation of antibiotic

SUMMARY:
The purpose of this study is to compare the effect of enhanced probiotic (EP, Live Rx) versus placebo (PL) on the incidence of Clostridium difficile associated diarrhea (CDAD) or antibiotic associated diarrhea (AAD) in hospitalized patients initiated on antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older admitted to SSH and prescribed antibiotics for an expected duration >3 days (may include patients on antibiotics prior to admission).

Exclusion Criteria:

* 1. History of chronic diarrhea illness (Irritable Bowel Disease (IBD), Irritable Bowel Syndrome (IBS), Celiac Disease, Chronic pancreatitis 2. Diarrhea at screening 3. Active Colitis of any etiology 4. History of colectomy 5. Regular consumption of probiotics within 72 hours 6. Unable to provide written consent 7. History of or active pancreatitis 8. Severe Sepsis or Septic Shock (sepsis with end organ failure e.g. renal failure, ARDS, MS changes and or meets criteria by n ational guideline, and or requiring vasopressors) 9. Hypersensitivity to any ingredient in probiotic product 10. Severe Immunosuppression (ANC <1000, AIDS/CD4 count <200 cells, cancer on active chemothereapy, h/o of solid or bone marrow transplant) 12. Acute burn injuries

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Incidence of Clostridium difficle associated diarrhea in patients randomized to Go Live Rx compared with those randomized to placebo | 60 days after hospitalization

SECONDARY OUTCOMES:
Incidence of Antibiotic associated diarrhea in patients randomized to Go Live Rx compared with those randomized to placebo | 60 Days after hospitalization